CLINICAL TRIAL: NCT05679076
Title: A Qualitative Study on the Pain and Quality of Life of Patients With Fabry Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1347
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry patients: Fabry patients

SUMMARY:
Background It is necessary to find out the difficulties experienced by patients with Fabry disease and their families, and to seek solutions for them. For this purpose, qualitative research with a patient-centered approach is useful.

Objectives The Objective of this study is to understand the various difficulties of patients with Fabry disease and to help them establish a comprehensive support system, medical, health, and welfare service system, and develop the direction and components of social and educational programs.

Methods The subjects of this study are patients who have been diagnosed with Fabry disease, and among them, are selected considering the selection and exclusion criteria, confirm consent for participation in the study after sufficient explanation, and then enroll. The target number of subjects is 10 people. Subjects who consented to the study had an in-depth interview centered on the in-depth interview questionnaire through the HA Research Institute, a specialized institution.

* The principle of saturation is observed by conducting 3 interviews per research subject.
* The duration of each interview per research subject is 50 to 60 minutes.
* All dictations of the research subjects were recorded with prior consent and then transcribed into a written copy.
* For 3 interviews, the number of interviews can be reduced to 1 or 2 by extending the interview time according to the research subject's request.
* As for the place of interview, the research counseling room at Severance Cardiovascular Hospital or the in-depth interview room in the HA Research Institute can be used, and the interview can be conducted at other places desired by the research subject at the request of the research subject.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have delayed diagnosis of Fabry disease or have experienced treatment refusal.
2. Subjects who have been diagnosed with Fabry name for more than 3 years or who have been treated for more than 1 year
3. Adults between the ages of 19 and 70 who have the ability to consent to participate in the research (excluding those subject to adult guardianship) and have the cognitive ability to dictate their experiences
4. Subjects who have experienced disadvantages and support in health-related quality of life, academic, job, family, social, and heterosexual relationships due to Fabry disease
5. Subjects who voluntarily gave written consent after hearing the explanation of the purpose and method of this clinical study

Exclusion Criteria:

1. Subjects who, in the opinion of the researcher, are unlikely to complete the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fabry patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-05-12 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Identify negative problems experienced by patients with Fabry disease | up to 5 months
Check the quality of life of patients with Fabry disease | up to 5 months
Identifying the structural causes of policies for patients with Fabry disease | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Geu-Ru Hong, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No